CLINICAL TRIAL: NCT00000681
Title: A Phase I Study of the Combination of Recombinant GM-CSF, AZT, and Chemotherapy (ABV) (Adriamycin, Bleomycin, Vincristine) in AIDS and Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 094; 11069 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Vincristine; Doxorubicin; Drug Evaluation; Drug Therapy, Combination; Granulocyte-Macrophage Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; Zidovudine; Bleomycin
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Bleomycin; Vincristine; Doxorubicin; Zidovudine; sargramostim

INTERVENTIONS:
Drug: Bleomycin sulfate
Drug: Vincristine sulfate
Drug: Doxorubicin hydrochloride
Drug: Zidovudine
Drug: Sargramostim

SUMMARY:
To determine the safety as well as the most effective dose of sargramostim (GM-CSF; granulocyte-macrophage colony stimulating factor) that will prevent the side effects caused by the combined use of zidovudine (AZT) and various doses of cancer-fighting drugs (doxorubicin, bleomycin, and vincristine) in AIDS patients with Kaposi's sarcoma (KS).

Patients included in this study have KS, which is a type of cancer that occurs in nearly 20 percent of patients with AIDS. AIDS patients with extensive KS require treatment with effective cytotoxic (anti-cancer) agents to reduce the tumor size and with antiretroviral agents such as AZT to prevent or ameliorate the development of opportunistic infections. Due to the significant toxic effect of both cytotoxic and antiviral agents on the bone marrow where new blood cells are generated, the combination of these agents is expected to result in complications such as granulocytopenia (very low granulocyte counts). Hematopoietic growth factors such as GM-CSF may reduce the severity and duration of marrow suppression. This may improve survival. Clinical trials of GM-CSF in HIV infected individuals with or without granulocytopenia have shown that the progenitor cells (early blood cells) are responsive to GM-CSF.

DETAILED DESCRIPTION:
Patients included in this study have KS, which is a type of cancer that occurs in nearly 20 percent of patients with AIDS. AIDS patients with extensive KS require treatment with effective cytotoxic (anti-cancer) agents to reduce the tumor size and with antiretroviral agents such as AZT to prevent or ameliorate the development of opportunistic infections. Due to the significant toxic effect of both cytotoxic and antiviral agents on the bone marrow where new blood cells are generated, the combination of these agents is expected to result in complications such as granulocytopenia (very low granulocyte counts). Hematopoietic growth factors such as GM-CSF may reduce the severity and duration of marrow suppression. This may improve survival. Clinical trials of GM-CSF in HIV infected individuals with or without granulocytopenia have shown that the progenitor cells (early blood cells) are responsive to GM-CSF.

AMENDED 910222 Due to continued concerns about GM-CSF toxicities seen in the 5 mcg/kg GM-CSF with 20 mg/m2 adriamycin/BV/AZT cohort, the GM-CSF dose in this study has been reduced while the adriamycin dose escalation will continue.

AMENDED 900430 Dosages for AZT and GM-CSF changed to reflect ongoing results. Original design: Patients receive the combination of AZT, antineoplastic chemotherapy, and GM-CSF in groups of three patients each. The first group receives baseline doses, and if the treatment is well tolerated, the subsequent groups of patients receive higher doses of the chemotherapy, in which the dose of doxorubicin is increased while bleomycin, vincristine, and AZT doses remain fixed throughout the study. The dose of all drugs remains fixed for a given patient. The anticancer drugs are given intravenously every 2 weeks. AZT is given every 4 hours by mouth. GM-CSF is self-injected subcutaneously every day from day 2 - day 12 of each treatment cycle. Patients repeat the chemotherapy every 2 weeks, for a maximum of seven cycles, with AZT being given continuously. When the maximum tolerated dose (MTD) of chemotherapy combined with GM-CSF is determined, the next phase of the study begins. Again the dose of chemotherapy is increased in groups of patients, but the every-day dose of GM-CSF is increased. Again, these chemotherapy cycles are repeated every 2 weeks up to a maximum of seven cycles. Patients receive physician examination and laboratory tests every week during the study and again at 4 weeks after the study. AMENDED: Dosages for AZT and GM-CSF have been changed to reflect ongoing results.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Non-steroidal agents such as acetaminophen for drug-related fevers.
* Pentamidine inhalation prophylaxis for Pneumocystis carinii pneumonia (PCP) in patients with a prior history or a T4 count < 200 cells/mm3.
* Antiemetics for nausea, vomiting.
* Symptomatic treatment for grades 1 and 2 oral toxicity.
* Toxicity grades according to NIAID Recommendations for Grading Acute and Subacute Toxic Effects (Adults).

Patients must have newly diagnosed biopsy-proven advanced AIDS-related Kaposi's sarcoma.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Systemic steroids for > 1 week in any 30 days.
* All known marrow-suppressive agents.
* Any other investigational drugs.

Patients will be excluded from the study for the following reasons:

* The presence of other active malignancies except basal cell carcinoma of the skin and in situ uterine cancer.
* Alteration of mental status that may not permit compliance with the protocol.
* Symptomatic sensory or motor neuropathy.
* History of myocardial infarction or significant arrhythmias.
* Class III/IV functional capacity in cardiac patients.

Prior Medication:

Excluded:

* Cytotoxic chemotherapy.

Excluded within 1 week of study entry:

* Therapy for Kaposi's sarcoma, including interferons, immunomodulators, antiretroviral agents.

Patients may not have any of the following diseases or symptoms:

* Allergy to bleomycin.
* The presence of other active malignancies except basal cell carcinoma of the skin and in situ uterine cancer.
* Alteration of mental status that may not permit compliance with the protocol.
* Symptomatic sensory or motor neuropathy.
* History of myocardial infarction or significant arrhythmias.
* Class III/IV functional capacity in cardiac patients.
* Concurrent serious infections, such as Pneumocystis carinii pneumonia (PCP), toxoplasma brain abscess, cytomegalovirus (CMV) retinitis or colitis, cryptococcal meningitis, and symptomatic Mycobacterium avium- intracellulare (MAI).

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Study Completion 1993-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gill PS, Study Chair; Miles S, Study Chair
Locations (5):
- United States (5):
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Pitt CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Gill PS, Bernstein-Singer M, Espina BM, Rarick M, Magy F, Montgomery T, Berry MS, Levine A. Adriamycin, bleomycin and vincristine chemotherapy with recombinant granulocyte-macrophage colony-stimulating factor in the treatment of AIDS-related Kaposi's sarcoma. AIDS. 1992 Dec;6(12):1477-81. doi: 10.1097/00002030-199212000-00009. PMID 1283520